CLINICAL TRIAL: NCT02668458
Title: Comparison of Pre-oxygenation by Non-invasive Ventilation With High-flow Nasal Oxygen Therapy for Intubation of Intensive Care Patients in Cases of Acute Respiratory Failure: A Prospective, Randomized, Controlled Study (FLORALI 2)
Brief Title: Comparison of Pre-oxygenation of NIV and HFNC Therapy for Intubation of ICU Patients With Acute Respiratory Failure
Acronym: FLORALI2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLORALI 2
Record Dates: First submitted 2016-01-19; First posted 2016-01-29 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Acute Respiratory Failure; Intratracheal Intubation
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NIV (Experimental): NIV group, preoxygenation by NIV: pressure support set for an exhaled tidal volume of 6-8 ml / kg of ideal body weight, PEEP of 5 cm H2O and FiO2 at 100%.
  Interventions: Procedure: Noninvasive ventilation
- HFNC (Active Comparator): High-flow nasal canula oxygen therapy. NHFC group, preoxygenation by NHFC: oxygen flow rate of 60 L / min and 100% FiO2
  Interventions: Procedure: High Flow nasal canula oxygen therapy

INTERVENTIONS:
Procedure: High Flow nasal canula oxygen therapy — Pre-oxygenation with high-flow nasal canula oxygen therapy
  Arms: HFNC
Procedure: Noninvasive ventilation — Pre-oxygenation with non-invasive ventilation
  Arms: NIV

SUMMARY:
The aim of the study is to evaluate the incidence of severe hypoxemia episodes during the intubation procedure with two methods of pre-oxygenation:

1. NIV (Non Invasive Ventilation)
2. HFNC (High-flow nasal canula oxygen therapy)

DETAILED DESCRIPTION:
Design:

Clinical randomized, open, multicenter, comparative trial, with parallel groups aimed at evaluating a medical device.

Selection of patients admitted to the ICU for acute respiratory failure, requiring endotracheal intubation.

Randomized study, inclusion in two groups: NIV or HFNC.

Experimental group:

NHFC group, preoxygenation by NHFC: oxygen flow rate of 60 L / min and 100% FiO2.

Control group:

NIV group, preoxygenation by NIV: pressure support set for an exhaled tidal volume of 6-8 ml / kg of ideal body weight, PEEP of 5 cm H2O and FiO2 at 100%.

Duration of participation of each patient: 28 days

ELIGIBILITY:
Main inclusion Criteria:

* acute hypoxemic respiratory failure requiring endotracheal intubation

Main exclusion Criteria:

* coma
* NIV contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Severe desaturation as defined by a pulse oxymetry below 80% | through five minutes after preoxygenation period
  drop below 80% of pulse oxymetry measurement

CONTACTS AND LOCATIONS:
Locations (27):
- France (27):
  - CHU Angers, Angers
  - CHU La cavale Blanche, Brest
  - CHU louis MOURIER, Colombes
  - Chu Mondor, Créteil
  - CHU Dijon, Dijon
  - CH Vendée, La Roche/Yon
  - CH La Rochelle, La Rochelle
  - CHU Lille, Lille
  - Limoges University Hospital, Limoges
  - CH St Joseph St Luc, Lyon
  - Chu E. Herriot, Lyon
  - LYON Sud, Lyon
  - CHU marseille, Marseille
  - CH, Montauban
  - CHU Lapeyronie, Montpellier
  - Hopital de l'Archet, Nice
  - CHU La Source, Orléans
  - Chu Cochin, Paris
  - CHU La Pitié Salpétrière, Paris
  - Chu Tenon, Paris
  - CHU Guadeloupe, Pointe à Pitre
  - CHU Poitiers, Poitiers
  - University Hospital of Poitiers, Poitiers
  - Hôpital C. NICOLLE, Rouen
  - CHU Strasbourg, Strasbourg
  - Hôpital FOCH, Suresnes
  - Chu Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez M, Ragot S, Coudroy R, Quenot JP, Vignon P, Forel JM, Demoule A, Mira JP, Ricard JD, Nseir S, Colin G, Pons B, Danin PE, Devaquet J, Prat G, Merdji H, Petitpas F, Vivier E, Mekontso-Dessap A, Nay MA, Asfar P, Dellamonica J, Argaud L, Ehrmann S, Fartoukh M, Girault C, Robert R, Thille AW, Frat JP; REVA Network. Noninvasive ventilation vs. high-flow nasal cannula oxygen for preoxygenation before intubation in patients with obesity: a post hoc analysis of a randomized controlled trial. Ann Intensive Care. 2021 Jul 22;11(1):114. doi: 10.1186/s13613-021-00892-8. PMID 34292408
- [Derived] Frat JP, Ricard JD, Quenot JP, Pichon N, Demoule A, Forel JM, Mira JP, Coudroy R, Berquier G, Voisin B, Colin G, Pons B, Danin PE, Devaquet J, Prat G, Clere-Jehl R, Petitpas F, Vivier E, Razazi K, Nay MA, Souday V, Dellamonica J, Argaud L, Ehrmann S, Gibelin A, Girault C, Andreu P, Vignon P, Dangers L, Ragot S, Thille AW; FLORALI-2 study group; REVA network. Non-invasive ventilation versus high-flow nasal cannula oxygen therapy with apnoeic oxygenation for preoxygenation before intubation of patients with acute hypoxaemic respiratory failure: a randomised, multicentre, open-label trial. Lancet Respir Med. 2019 Apr;7(4):303-312. doi: 10.1016/S2213-2600(19)30048-7. Epub 2019 Mar 18. PMID 30898520
- [Derived] Frat JP, Ricard JD, Coudroy R, Robert R, Ragot S, Thille AW; on-behalf-of REVA network. Preoxygenation with non-invasive ventilation versus high-flow nasal cannula oxygen therapy for intubation of patients with acute hypoxaemic respiratory failure in ICU: the prospective randomised controlled FLORALI-2 study protocol. BMJ Open. 2017 Dec 22;7(12):e018611. doi: 10.1136/bmjopen-2017-018611. PMID 29275345